CLINICAL TRIAL: NCT03859167
Title: SLAVSME - Study of the Loss of AV Synchrony at Maximum Exercise
Brief Title: Study of the Loss of AV Synchrony at Maximum Exercise
Acronym: SLAVSME
Status: Terminated | Type: Observational
Why Stopped: No Enrollments after COVID
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Jay Montgomery, Assistant Professor, Vanderbilt University Medical Center
Other Study IDs: 190470
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Exercise; Pacemaker; Blood Pressure
MeSH Terms: conditions — Motor Activity | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with AV block with pacemaker: Participants will have a stress test, and results will be collected and recorded.
  Interventions: Other: Stress Test

INTERVENTIONS:
Other: Stress Test — Participants will reach maximum exercise on a treadmill and results will be collected and recorded.

SUMMARY:
Investigators will identify a group of patients with complete heart block and a dual chamber pacemaker who will be expected to be able to exercise on a treadmill. Investigators will utilize symptom logs, cuff and continuous blood pressure monitoring. It is planned to study the symptomatic impact of loss of AV synchrony at significant levels of exercise.

ELIGIBILITY:
Inclusion Criteria:

* Complete AV Block
* Age less than 60
* Easily programmable dual chamber pacemaker

Exclusion Criteria:

* Age > 60
* Significant Heart Failure
* Significant angina
* History of claudication
* Significant orthopedic issues
* Evidence of sinus node dysfunction
* Taking beta blockers or non-dihydropyridine calcium channel blockers

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: patients from cardiology clinic
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
The number of participants with Loss of AV synchrony at maximum exercise | Baseline to end of stress test approximately 60 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Jay A. Montgomery, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided